CLINICAL TRIAL: NCT01021527
Title: A Randomized, 4-Period Study to Assess the Effects of Exenatide on Insulin Secretion Rates Using a Graded Infusion of Intravenous Glucose
Brief Title: A Study to Assess the Effects of Exenatide on Insulin Secretion Rates Using a Graded Infusion of Intravenous Glucose (0000-099)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-099; 099; 2009_697
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence 1 (Experimental): A-B-C-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion
- Treatment Sequence 2 (Experimental): B-C-A-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion
- Treatment Sequence 3 (Experimental): C-A-B-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion
- Treatment Sequence 4 (Experimental): A-C-B-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion
- Treatment Sequence 5 (Experimental): B-A-C-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion
- Treatment Sequence 6 (Experimental): C-B-A-C
  Interventions: Other: Comparator: Treatment A; Drug: Comparator: Treatment B; Drug: Comparator: Treatment C; Procedure: Comparator: graded glucose infusion

INTERVENTIONS:
Other: Comparator: Treatment A — No Treatment
Drug: Comparator: Treatment B — single dose administration of exenatide 5ug by subcutaneous injection
Drug: Comparator: Treatment C — single dose administration of exenatide 10ug by subcutaneous injection
Procedure: Comparator: graded glucose infusion — A stepwise graded infusion of glucose (20% dextrose [D20]) with a stable rate of infusion maintained for 40 minutes for each of 5 steps, with steps at 2,4,6,8 and 12 mg/kg/min. Infusion will be performed during each of the 4 treatment periods.

SUMMARY:
A four-period study to evaluate if the grade glucose infusion procedure will be able to detect an increase in beta-cell glucose sensitivity from exenatide compared to no treatment in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a non-smoker

Exclusion Criteria:

* Subject has irritable bowel disease
* Subject has a history of cancer
* Subject has a history of hypertension requiring treatment
* Subject is unable to refrain from the use of any prescription or non-prescription medication
* Subject consumes excessive amounts of alcohol or caffeine
* Subject has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
beta-cell glucose sensitivity (slope of the relationship between insulin secretion rate and glucose) | 0-160 minutes after start of infusion

SECONDARY OUTCOMES:
safety and tolerability of a graded glucose infusion procedure measured by the number of clinical adverse experiences | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC